CLINICAL TRIAL: NCT04731441
Title: Exercise Intervention Prior to CRS-HIPEC: Feasibility & Impact
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling and we lost exercise specialist
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Colette Pameijer, Professor, Department of Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015358
Record Dates: First submitted 2021-01-15; First posted 2021-02-01 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Colon Cancer; Ovarian Cancer; GI Cancer; Gynecologic Cancer
Keywords: HIPEC; CRS; Prehabilitation; Exercise
MeSH Terms: conditions — Colonic Neoplasms; Ovarian Neoplasms; Gastrointestinal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects will be partially randomized to 1 of 2 treatment arms. Sarcopenia will be measured at baseline but is not a criterion for enrollment. Sarcopenic patients will all be in the intervention arm and receive the prehab exercise program. Non-sarcopenic patients will be randomized to the intervention arm or the control arm. The allocation scheme for non-sarcopenic subjects will be made with a computerized random number generator. This will take place the day of consent and subjects will be notified in person by the research assistant before the end of their visit with the surgeon.
  After randomization, subjects will proceed with a baseline assessment to obtain basic demographics, muscle strength, endurance performance, physical functioning, and physical activity. The subject will then proceed with 6 weeks of participating in the control or intervention arm, followed by surgery and a post-operative assessment. After the post-operative assessment, study is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Exercise Program Subjects randomized to the intervention arm should have 6 weeks of home exercise prior to surgery, with a minimum of 5 weeks and not more than 7 weeks. The program will begin with an exercise consultation appointment with a certified fitness professional. During this consultation participants will receive an exercise manual for individualized home-based exercise and a practical introduction by an exercise and cancer specialist. PowerBlock adjustable dumbbells will be used for resistance training exercises and walking or jogging will be the primary type of aerobic training. The current program design was developed and successfully used with women with breast cancer. Thus, some components may need modification for this group of patients with advanced GI cancer.
  Interventions: Behavioral: Home-based Exercise Program Prior to CRS-HIPEC
- Education Group (Active Comparator): Subjects randomized to the control arm will receive education and a handbook on the benefits of exercise and will be encouraged to have adequate protein in their diet and provided with the list of high protein foods and nutritional information. These subjects will undergo the same assessments as the intervention arm at all time points. Control subjects will be offered a 6-week home exercise program 3 months after CRS/HIPEC. Results and outcomes will not be recorded.
  Interventions: Behavioral: Exercise Education

INTERVENTIONS:
Behavioral: Home-based Exercise Program Prior to CRS-HIPEC — Exercise Program Subjects randomized to the intervention arm should have 6 weeks of home exercise prior to surgery, with a minimum of 5 weeks and not more than 7 weeks. The program will begin with an exercise consultation appointment with a certified fitness professional. During this consultation participants will receive an exercise manual for individualized home-based exercise and a practical introduction by an exercise and cancer specialist. PowerBlock adjustable dumbbells will be used for resistance training exercises and walking or jogging will be the primary type of aerobic training. The current program design was developed and successfully used with women with breast cancer. Thus, some components may need modification for this group of patients with advanced GI cancer.
  Arms: Exercise Group
Behavioral: Exercise Education — Control arm: Subjects randomized to the control arm will receive education and a handbook on the benefits of exercise and will be encouraged to have adequate protein in their diet and provided with the list of high protein foods and nutritional information. These subjects will undergo the same assessments as the intervention arm at all time points. Control subjects will be offered a 6-week home exercise program 3 months after CRS/HIPEC, as described in sections 7.2.1-7.2.3. Results and outcomes will not be recorded.
  Arms: Education Group

SUMMARY:
Our objective is to initiate an exercise program for patients with advanced GI or Gyn cancer, as prehabilitation prior to surgery. The objective of the prehabilitation program is to reduce complication rates and improve the length and quality of survival for patients with abdominal cancer. The prehabilitation program will be offered to patients who are eligible for and consent to cytoreductive surgery (CRS) and heated intraperitoneal chemotherapy (HIPEC)

DETAILED DESCRIPTION:
Our objective is to assess the feasibility and impact of implementing an exercise program for patients with advanced GI or Gyn cancer, as prehabilitation prior to surgery. The objective of the prehabilitation program is to reduce complication rates and improve the length and quality of survival for patients with abdominal cancer. The prehabilitation program will be offered to patients who are eligible for and consent to cytoreductive surgery (CRS) and heated intraperitoneal chemotherapy (HIPEC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with peritoneal metastasis from appendix, colon, small bowel, endometrium, ovary or any other GI or Gyn primary tumor
* Patients should be eligible for and consent to surgery with the intention of performing CRS / HIPEC at Penn State Hershey Medical Center. Eligibility for CRS/HIPEC is a clinical determination based on a combination of factors including radiographic extent of disease, tumor histology and medical fitness for surgery
* Subjects who are explored but found to be unresectable will be included.
* Male or female.
* Patients should be age 18 or above.
* Surgery is planned for not less than 6 weeks and no more than 10 weeks from consultation

Exclusion Criteria:

* Patients who do not consent to surgery.
* Patients who require urgent surgery, sooner than 6 weeks
* Patients receiving neoadjuvant chemotherapy, with no surgical date planned before 10 weeks from consultation. These patients can be enrolled at the time of the follow-up visit, as long as they meet above criteria
* Patients not fluent in English
* Pregnant women
* Prisoners
* Patients with Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptability | 1 year
  Rate of enrollment into this trial
Feasibility of doing exercises | 2 months
  The percent of exercises completed by subjects

SECONDARY OUTCOMES:
30-day Complication | 1 month
  • To assess the 30-day rate of complications after prehabilitation and CRS/HIPEC. The rate of complication after CRS/HIPEC is well described in the literature and established in our patient population at Penn State Cancer Institute. Infectious and non-infectious complications and length of stay will be collected
Quality of Life after CRS-HIPEC | 1 year
  • To monitor quality of life after prehabilitation and CRS/HIPEC. Quality of life (QOL) after CRS/HIPEC is well described in the literature and was assessed in our patients in a pilot study that is nearly completed. Patient-Reported Outcomes Measurement Information System (PROMIS) T-Scores for Physical Function will be obtained, scores ranging from 20-80, with higher scores reflecting higher physical function.
  To assess the effects of prehabilitation and CRS/HIPEC on muscle mass. Muscle mass at the level of L3 on cross-sectional imaging will be measured for all subjects at baseline, to determine the presence of sarcopenia. Muscle mass will be measured again after CRS/HIPEC. Changes in muscle mass after CRS/HIPEC are unknown, and the effect of a prehabilitation program in this patient population are also unknown. The results will serve as preliminary data for a future, larger study in this population with more specific hypotheses.

CONTACTS AND LOCATIONS:
Overall Officials: Colette R Pameijer, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Non-applicable